CLINICAL TRIAL: NCT05960305
Title: A Multi-Site Randomized Actual Use Study of Electronic Nicotine Delivery System (P12) Products Among Current U.S. Adult Smokers to Assess the Relative Impact of Availability and Use of Different E-liquid Flavors on Changes in Cigarette Consumption
Brief Title: CSD201204 An Actual Use Study of P12 Electronic Nicotine Delivery System Among U.S. Adult Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CSD201204
Record Dates: First submitted 2023-07-10; First posted 2023-07-25 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Smoking, Tobacco
Keywords: Smoking, Tobacco Use, Tobacco Smoking
MeSH Terms: conditions — Tobacco Smoking; Smoking; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tobacco Flavor (Active Comparator): Can choose between 2 different tobacco flavor variants at 2 different nicotine levels (1.5% and 5%)
  Interventions: Other: P1213416; Other: P1213422; Other: P1213716; Other: P1213722
- Menthol Flavor (Active Comparator): Can choose between 2 different menthol flavor variants at 2 different nicotine levels (1.5% and 5%)
  Interventions: Other: P1211216; Other: P1211222; Other: P1213616; Other: P1213622
- NTNM Flavor (Active Comparator): Can choose between 2 different non tobacco/non menthol flavor variants at 2 different nicotine levels (1.5% and 5%)
  Interventions: Other: P1213816; Other: P1213822; Other: P1211916; Other: P1211922

INTERVENTIONS:
Other: P1213416 — Tobacco Flavor
  Arms: Tobacco Flavor
Other: P1213422 — Tobacco Flavor
  Arms: Tobacco Flavor
Other: P1213716 — Tobacco Flavor
  Arms: Tobacco Flavor
Other: P1213722 — Tobacco Flavor
  Arms: Tobacco Flavor
Other: P1211216 — Menthol Flavor
  Arms: Menthol Flavor
Other: P1211222 — Menthol Flavor
  Arms: Menthol Flavor
Other: P1213616 — Menthol Flavor
  Arms: Menthol Flavor
Other: P1213622 — Menthol Flavor
  Arms: Menthol Flavor
Other: P1213816 — NTNM Flavor
  Arms: NTNM Flavor
Other: P1213822 — NTNM Flavor
  Arms: NTNM Flavor
Other: P1211916 — NTNM Flavor
  Arms: NTNM Flavor
Other: P1211922 — NTNM Flavor
  Arms: NTNM Flavor

SUMMARY:
The purpose of this Actual Use Study (AUS) is to investigate how United States (US) adult tobacco consumers 21 to 60 years of age, inclusive, who are regular smokers (≥5 cigarettes/day on at least 20 of the past 30 days) will use the Cartridge-based ENDS investigational products (Study IP) over a 6-week Actual Use Period (AUP) in their real-life/naturalistic environments. Subjects will be able to choose freely among the Study IP available in one of the three study arms to which they are randomly assigned. The three study arms are organized by Study IP flavor categories: tobacco, menthol, and non-tobacco-non-menthol (NTNM). Subjects will self-report their ad libitum use of the Study IP as well as use of Combustible Cigarettes (CC) and any other tobacco- and nicotine-containing product (TNP) on a daily basis using an electronic diary (eDiary).

DETAILED DESCRIPTION:
The AUS is a multi-site, open-label, randomized, three-arm, 8-week, prospective observational study to be conducted at multiple sites geographically dispersed within the U.S.. Adult tobacco consumers 21 to 60 years of age (inclusive) who smoked on at least 20 of the past 30 days and smoked at least 5 CPD on the days they smoked will be provided the Study IP for ad libitum use over a 6-week Actual Use Period (AUP) in their real-life/naturalistic environments. Subject-reported consumption of the Study IP, Combustible cigarettes, and other TNPs will be assessed (including, but not limited to, ENDS, smokeless tobacco, and other combustible tobacco products).

The study includes pre-screening, a screening and enrollment visit (SEV), a baseline assessment period (BAP), an observational actual use period (AUP), and a close out period (COP). Following the recruitment period, the study duration per enrolled subject will be approximately eight (8) weeks. Following the administration of a Baseline Assessment Questionnaire (BAQ) at the SEV, use of Combustible Cigarettes and other TNP will be self-reported using an eDiary during the 1-week BAP.

At SEV, subjects will be asked to indicate their likelihood to use each Study IP flavor variant across the three study arms. Subjects who indicate an interest in using at least one of the two flavors per arm for all three arms will be enrolled into the study and randomized into one of the three arms prior to completion of BAQ.

The Study IP evaluated in this study will include the Power Unit and 12 cartridge variants (six flavor variants in two nicotine concentrations, 1.5% and 5%). In each arm, four variants (two flavor variants in two nicotine concentrations) will be available for choice. Subjects will be shown the Study IP (power unit, charging cord and all 12 flavor cartridges), user guide and handout marketing materials (MM) at SEV prior to study arm assignment. MM (poster) of Study IP in all three arms will be present at SEV and only arm-specific MM will be present at all subsequent site visits. Subjects will be first dispensed the power unit and preferred Study IP variants (i.e., specific flavor and nicotine concentrations) available within their assigned study arm during SV1 and a handout MM will be given to the subjects to take home at SV1.

Starting at SV1, enrolled subjects will be able to select Study IP for use during the AUP from the Study IP available in their assigned study arm. Subjects will be instructed not to use ENDS other than the Study IP provided by the study site for the duration of the AUP in the ICF. However, if subjects report other ENDS use in the eDiary, this will not lead to study discontinuation. Subjects can use the Study IP and other TNP including Combustible Cigarettes ad libitum during the AUP and will self-report product use on a daily basis via an eDiary over the 6-week AUP. Throughout the AUP, a toll-free Hotline will be available for subjects to report potential product-related adverse health experiences, pregnancy, and/or product quality complaints.

Subjects will return to the study site three additional times (SV2, SV3, and SV4) for an interview to review eDiary compliance, complete additional questionnaires, return unused Study IP, and receive additional Study IP (SV2 and SV3, as needed). At SV4, subjects will complete an End of Study Questionnaire (ESQ). The COP will allow for reporting study queries to the sites, along with possible adverse health experiences to the toll-free Hotline after SV4.

Subjects will be presented with hard-copy marketing material (MM) at the SEV for all Study IP variants in all three study arms. Consistent with typical consumer marketing practices, representative point of sale (POS) MM will be present during subject interactions at the SEV and SVs (e.g., product poster). At SV1-SV4, enrolled subjects will only be exposed to MM relating to the Study IP variants for the respective study arm they are randomized into.

ELIGIBILITY:
Inclusion Criteria:

* 1. Generally healthy adult males or females, 21-60 years old, inclusive, verified with government-issued photo ID.

  2. Must be a current smoker of manufactured menthol and/or non-menthol cigarettes, has smoked at least 100 cigarettes in their lifetime, and smoked on at least 20 days out of the past 30 days.

  3. Smokes, on average, ≥ 5 Combustible cigarettes per day (CPD) on days when cigarettes are smoked (in the past 30 days).

  4. Must indicate "an intention to use" (6 or higher on a 10-point Likert scale) for at least one Study IP flavor per arm across all three study arms after a brief review of the products and related information (i.e. User Guide and Handout MM) at the SEV.

  5. Has not participated in any tobacco-, ENDS-, or nicotine-related research within 1 month of screening.

  6. Must sign the Informed Consent Forms (ICFs) and thereby agree to participate in the 8-week study, comply with all study requirements, including eDiary reporting procedures and completion of questionnaires/eDiary in English, and agree that the Study IP received are for their own personal use and will not be shared with others.

Exclusion Criteria:

* 1. Self-reports as currently quitting or intending to quit within the next 3 months all tobacco or nicotine product use ("currently" is defined as within [≤] 30 days prior to pre-screening).

  2. Currently a regular ENDS user (using ENDS >3 days per week, in the past 30 days), based on self-report.

  3. Female subjects who are pregnant or breastfeeding or planning to become pregnant or start breastfeeding within the next 6 months based on self-report.

  4. Female subjects who state they are not using adequate methods to prevent pregnancy.

  5. Female subjects (as assigned at birth) who do not have a definitive negative pregnancy test result at SEV.

  6. Self-reports "poor" physical health

  7. Self-reports "poor" mental health

  8. Employees of a company that manufactures tobacco or ENDS products.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1845 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-28 (Actual)

PRIMARY OUTCOMES:
Number and proportion of subjects who reduce their cigarettes per day (CPD). | 6 weeks
  Number and proportion of subjects who reduce their cigarettes per day (CPD) consumption by at least 50% at Week 6 compared to baseline among all subjects who complete the study.
CPD mean percent reduction | 6 weeks
  CPD mean percent reduction at Week 6 compared to baseline among all subjects who complete the study.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Jordan, PhD, Study Director — RAIS
Locations (12):
- United States (12):
  - Sago Phoenix, Phoenix, Arizona
  - Non Sago Ft Lauderdale, Fort Lauderdale, Florida
  - SAGO Orlando, Orlando, Florida
  - Non Sago Tampa, Tampa, Florida
  - Sago Atlanta, Atlanta, Georgia
  - Sago St. Louis, St Louis, Missouri
  - Non-Sago Las Vegas, Las Vegas, Nevada
  - Sago Philadelphia, Philadelphia, Pennsylvania
  - Sago Nashville, Nashville, Tennessee
  - Sago Dallas, Dallas, Texas
  - Sago Houston, Houston, Texas
  - Non Sago San Anotonio, San Antonio, Texas